CLINICAL TRIAL: NCT01711853
Title: An Exploratory Study to Investigate the Pharmacokinetics and Effects of DABIgatran Etexilate in Patients With Stable Severe RENAL Disease: DabiRenal
Brief Title: Study to Evaluate the Pharmacokinetics and Pharmacodynamics of Dabigatran Etexilate in Patients With Stable Severe Renal Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1160.166; 2011-003081-32 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-10-19; First posted 2012-10-22 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Dabigatran

ARMS (1):
- Dabigatran Etexilate (Experimental): patient to receive a capsule containing 75 mg of dabigatran etexilate
  Interventions: Drug: Dabigatran Etexilate

INTERVENTIONS:
Drug: Dabigatran Etexilate — Dabigatran Etexilate 75mg twice daily

SUMMARY:
The study to be conducted is a prospective, open label trial. It is designed to evaluate the pharmacokinetic/pharmacodynamic and coagulation parameters and safety of dabigatran etexilate in patients with chronic kidney disease.

ELIGIBILITY:
Inclusion criteria:

1. Male and female patients aged 18 years and older
2. Impaired renal function defined as a stable Cockcroft-Gault and/or actual creatinine clearance between 15-30 ml/min over the last 3 months before study participation.
3. The single use of either aspirin or Vitamin K Antagonists
4. Provision of informed consent.

Exclusion criteria:

1. Unstable renal function and Creatinin Clearance <15mL/min
2. Patients treated with two or more platelet aggregation inhibitors
3. Use of or indication for therapeutic heparin
4. Patients with prosthetic heart valves
5. Haemorrhagic disorder or bleeding diathesis
6. Platelet count <100 109/L) at screening or during the last 30 days before screening.
7. Participation in another drug trial in the last 30 days before screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1160.166.31001 Boehringer Ingelheim Investigational Site, Leiden, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Dabigatran 75 mg: Oral administration of 1 capsule of Dabigatran etexilate 75 mg twice daily
Period: Overall Study
Arm/Group | Dabigatran 75 mg
Started | 19
Completed | 16
Not Completed | 3
Not completed — Not treated | 3

BASELINE CHARACTERISTICS:
Population: Treated set (TS) which included all patients who had taken at least 1 dose of trial medication.
Arm/Group | Dabigatran 75 mg
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Cmax,ss
Description: Maximum concentration of Dabigatran etexilate in plasma at steady state was measured.
  The samples for pharmacokinetics had to be taken from 30 min before drug administration up to 11 days after drug administration.
Time Frame: -0.5 hours (h), 0.5h, 1h, 2h, 3h, 4h, 6h, 8h, 12h, 23.5h, 47.5h, 71.5h, 95.5h, 119.5h, 155.5h, 167.5h, 168.5h, 169h, 170h, 171h, 172h, 174h, 176h, 179.5h, 180h, 192h, 216h, 240h
Population: Pharmacokinetic set (PKS) which included all treated subjects that provided at least 1 observation for at least 1 primary pharmacokinetic endpoint without important protocol violations with respect to the evaluation of the pharmacokinetic endpoints and with predose values not greater than 5% of Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran 75 mg
Number analyzed (Participants) | 15
ng/mL | 207 (53.9)
Statistical Analysis 1: Comparison: Dabigatran 75 mg; Patients were classified into groups for renal function based on the median values for renal function (1: ≤ median GFR (Glomerular filtration rate), 2: > median GFR). Median is calculated based on trial data of treated set; Test type: Superiority or Other; p = 0.5186, ANOVA; ANOVA model on the logarithmic scale; effects accounting for the following sources of variation: 'gender', 'age group', and 'renal function group'
Statistical Analysis 2: Comparison: Dabigatran 75 mg; Patients were classified into groups for renal function based on the median values for renal function (1: ≤ median age, 2: > median age). Median is calculated based on trial data of treated set; Test type: Superiority or Other; p = 0.9883, ANOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dabigatran 75 mg; Patients were classified based on the gender distribution; Test type: Superiority or Other; p = 0.7853, ANOVA; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: AUCtau,ss
Description: Area under the plasma concentration-time curve of the total dabigatran at steady state over a uniform dosing interval tau was measured.
  The samples for pharmacokinetics had to be taken from 30 min before drug administration up to 11 days after drug administration.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dabigatran 75 mg
Number analyzed (Participants) | 15
ng*h/mL | 2140 (51.9)
Statistical Analysis 1: Comparison: Dabigatran 75 mg; Patients were classified into groups for renal function based on the median values for renal function (1: ≤ median GFR, 2: > median GFR). Median is calculated based on trial data of treated set; Test type: Superiority or Other; p = 0.4692, ANOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Dabigatran 75 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.9734, ANOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Dabigatran 75 mg; Patients were classified based on the gender distribution; Test type: Superiority or Other; p = 0.9201, ANOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to Day 11
Arm/Group | Dabigatran 75 mg
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 6/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 75 mg (N=16)
Diarrhoea (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Nail injury (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Thrombophlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights